CLINICAL TRIAL: NCT03579212
Title: National, Multicentre, Prospective, Retrospective, Observational Study, to Evaluate the Performance of Y-STRUT® Medical Device to Strengthen Pre-fractural Tumour-induced Lesions at the Level of the Proximal Femur
Brief Title: Evaluation of the Performance of Y-STRUT® Medical Device to Strengthen Pre-fractural Tumour-induced Lesions at the Level of the Proximal Femur
Status: Terminated | Type: Observational
Why Stopped: EC withdrawal with termination of the NB contract
Sponsor: Hyprevention (Industry)
Responsible Party: Sponsor
Other Study IDs: HIPPON100
Record Dates: First submitted 2017-09-22; First posted 2018-07-06 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2020-06

CONDITIONS: Pathological Fracture of Hip; Bone Metastases
Keywords: Osteosynthesis; Prophylactic consolidation; Proximal femur

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Y-STRUT® (Hyprevention, Pessac, France) — The studied medical device consists of two components implanted in the proximal femur, combined with bone cement.

SUMMARY:
HIPPON 100 is a national, multicentre, prospective, retrospective, descriptive and non-interventional study, in patients having a Y-STRUT® medical device implanted to prevent a high risk of impending pathological fracture.

The primary objective of this study is to evaluate the performance of the studied medical device by measuring the frequency of patient with a fracture at the implantation site within 1 year after implantation.

A total of 100 patients from France will be enrolled (until November 2018) and followed up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old
* Patient with information form signed to participate in the study;
* Patient presenting a cancer with bone metastases at the level of the proximal femur and having a Y-STRUT® medical device implanted;
* Patient able to complete a questionnaire.

Exclusion Criteria:

* Patient who refuse to participate to this study;
* Patient already enrolled in a clinical study, excluding his participation to HIPPON100.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with a Y-STRUT® device to strengthen pre-fractural tumour-induced lesions at the level of the proximal femur.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Frequency of post-operative fracture [Performance of the device] | At 12 months
  Frequency of patient with a fracture at the implantation site

SECONDARY OUTCOMES:
Frequency of post-operative fracture [Performance of the device] | At 6 and 24 months
  Frequency of patient with a fracture at the implantation site
Pain [Tolerance of the device] | immediate post-op, and at 6, 12 and 24 months
  Self-evaluation of pain using VAS (Visual Analogue Scale), going from 0 (no pain) to 10 (maximum).
Resumption of weight-bearing [Tolerance of the device] | immediate post-op, and at 6, 12 and 24 months
  Assessment of resumption of weight-bearing (yes/no at each visit)
Quality of life [Tolerance of the device] | pre-operative, immediate post-op, and at 6, 12 and 24 months
  Assessment of the quality of life using EORTC QLQ-C15-PAL questionnaire: the European Organization for Research and Treatment of Cancer (EORTC) has developed the QLQ-C15-PAL questionnaire (quality of life questionnaire with 15 items), a short version of the QLQ-C30 for palliative (PAL) care. Scale ranges go from 15 (better) to 63 points (worse) at the maximum.
Recording of adverse events and device effects [Safety of the device] | At 6, 12 and 24 months
  Recording of the medical device vigilance: all serious adverse events, all adverse events linked to the device or the operative technique, and any other important event reported.
Surgical procedure duration [feasibility of the procedure] | At inclusion (day 1)
  Measuring mean/median intervention duration.
Hospitalisation duration [feasibility of the procedure] | At inclusion (day 1)
  Measuring mean/median hospitalisation duration.
Rates of complications [feasibility of the procedure] | At inclusion (day 1)
  Assessing types and frequencies of procedures complications.
Calculation of associated costs [Economic impact of the procedure] | At the end of the study (24 months from the last included patient)
  Evaluation of each cost associated with all the collected data linked to the procedure (implantation costs, hospitalisation costs, treatments for pain and other events). Then, the different costs are added together to determine the mean total cost of a procedure.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CHU Caen, Caen
  - Hôpital européen Georges-Pompidou, Paris
  - Hopital Tenon - AP-HP, Paris
  - CHU Toulouse, Toulouse